CLINICAL TRIAL: NCT02794285
Title: A Multicentre, Randomised, Double-blind, Placebo-Controlled Phase 3 Extension Study to Characterise the Long-term Safety and Tolerability of Anifrolumab in Adult Subjects With Active Systemic Lupus Erythematosus.
Brief Title: Long Term Safety of Anifrolumab in Adult Subjects With Active Systemic Lupus Erythematosus
Acronym: TULIP SLE LTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3461C00009
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Active Systemic Lupus Erythematosus
Keywords: Lupus Erythematosus, Systemic Autoimmune Diseases, Connective Tissue Diseases,Immune System Diseases
MeSH Terms: conditions — Connective Tissue Diseases; Immune System Diseases | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anifrolumab (Experimental): Anifrolumab
  Interventions: Biological: Anifrolumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Anifrolumab — Anifrolumab IV administration every 4 weeks from Week 0 to Week 152 for a total of 39 doses
  Arms: Anifrolumab
Drug: Placebo — Placebo IV administration every 4 weeks from Week 0 to Week 152 for a total of 39 doses
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterise long-term safety and tolerability of intravenous anifrolumab.

DETAILED DESCRIPTION:
This is a Phase 3, multicentre, multinational, randomised, double-blind, placebo-controlled extension study to characterising the long term safety and tolerability of of an intravenous treatment regimen of anifrolumab versus placebo in subjects with moderately to severely active systemic lupus erythematosus who completed a Phase 3 study (D3461C00004 or D3461C00005) through the 52-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have qualified for and received investigational product (anifrolumab or placebo) and completed the treatment period in Studies D3461C00004 or D3461C00005 (through Week 52)
2. Adequate peripheral venous access
3. Females with an intact cervix should have documentation of a Pap smear with no documented malignancy within 90 days before Day 1/Visit 1 or 30 days following Day 1/Visit 1. Since access to a Pap smear may vary by country, the Sponsor recommends that local guidelines for obtaining Pap smears in subjects who have received immunomodulators or immunosuppressive treatment be followed.
4. Meets the following TB criteria:

   1. Negative QuantiFERON®-TB Gold [QFT-G] test result for TB obtained from the study central laboratory at Week 52 of Studies D3461C00004 or D3461C00005; OR
   2. Newly positive QFT-G test result at Week 52 of Studies D3461C00004 or D3461C00005 from the study central laboratory. A chest x-ray must be performed. If the chest x-ray shows no evidence of active TB, and the subject has no symptoms or medical history consistent with active TB, the subject must have a retest. If the retest is positive, the subject must start on prophylaxis within 30 days of randomisation but prior to the second dose of investigational product (Visit 2/Week 4); OR
   3. Positive but not newly positive QFT-G test at Week 52 of Studies D3461C00004 or D3461C00005. The subject must have been diagnosed with latent TB and must have documentation confirming initiation of appropriate treatment OR initiate treatment for latent TB within 30 days of randomization, but prior to the second dose of investigational product administration (Visit 2/Week 4)
   4. Newly indeterminate (confirmed on retest unless prior positive QFT G was documented, along with completed treatment for latent TB) or indeterminate but not newly indeterminate QFT-G test result at Week 52 of Studies D3461C00004 or D3461C00005 from the study central laboratory with ongoing QFT-G testing for TB according to the Study Plan
5. In the opinion of the Investigator, subject must be able to comprehend the ICF and all protocol related assessments

Exclusion Criteria:

1. Receipt of any of the following within the last 60 days:

   1. Azathioprine >200 mg/day
   2. Mycophenolate mofetil >2.0 g/day /mycophenolic acid >1.44 g/day
   3. Oral, subcutaneous, or intramuscular methotrexate >25 mg/week
   4. Mizoribine >150 mg/day
2. Receipt of any investigational product (small molecule or biologic agent other than anifrolumab) within 4 weeks or 5 half-lives prior to Day 1/Visit 1, whichever is greater
3. Receipt of any of the following:

   1. Any live or attenuated vaccine within 8 weeks prior to Day 1/Visit 1 (administration of killed vaccines is acceptable, the Sponsor recommends Investigators ensure all subjects are up to date on required vaccinations, including influenza [inactivated/recombinant] vaccine prior to study entry)
   2. Bacillus Calmette-Guerin (BCG) vaccine between the end of Studies D3461C00004 or D3461C00005 and Day 1/Visit 1
4. Active severe SLE-driven renal or neuropsychiatric disease
5. Any underlying condition that predisposes the subject to infection, including history of/current human immunodeficiency virus (HIV) infection
6. Subjects with Hepatitis B core antibody (HBcAb) positivity at enrolment of Studies D3461C00004 or D3461C00005 will be tested every 3 months for Hepatitis B virus (HBV) DNA. To remain eligible in the LTE study, subject HBV DNA levels must remain below the lower limit of quantitation as per the central laboratory.
7. Opportunistic infection requiring hospitalisation or parenteral antimicrobial treatment within 3 years of Day 1/Visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kalunian, MD, Principal Investigator — University of California, San Diego; Raj Tummala, MD, Study Director — AstraZeneca
Locations (154):
- United States (53):
  - Research Site, Birmingham, Alabama
  - Research Site, El Cajon, California
  - Research Site, Hemet, California
  - Research Site, La Jolla, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, San Leandro, California
  - Research Site, Thousand Oaks, California
  - Research Site, Upland, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Brandon, Florida
  - Research Site, DeBary, Florida
  - Research Site, Miami, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Cumberland, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Nashua, New Hampshire
  - Research Site, Freehold, New Jersey
  - Research Site, Las Cruces, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Great Neck, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, North Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Stafford, Texas
  - Research Site, Spokane, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, San Miguel de Tucumán
- Australia (2):
  - Research Site, Fitzroy
  - Research Site, Kogarah
- Research Site, Plovdiv, Bulgaria
- Canada (2):
  - Research Site, Hamilton, Ontario
  - Research Site, Rimouski, Quebec
- Chile (3):
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Viña del Mar
- Colombia (3):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Medellín
- France (5):
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
- Germany (6):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Kirchheim
  - Research Site, Mainz Am Rhein
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Tel Aviv
- Japan (13):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kitakyushu-shi
  - Research Site, Kurashiki-shi
  - Research Site, Meguro-ku
  - Research Site, Nagasaki
  - Research Site, Omura-shi
  - Research Site, Sapporo
  - Research Site, Sasebo-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Klaipėda
- Mexico (6):
  - Research Site, Chihuahua City
  - Research Site, León
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, México
  - Research Site, San Luis Potosí City
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Poland (10):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Nadarzyn
  - Research Site, Starachowice
  - Research Site, Szczecin
  - Research Site, Ustroń
  - Research Site, Warsaw
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Galati
  - Research Site, Târgu Mureş
- Russia (4):
  - Research Site, Smolensk
  - Research Site, Tolyatti
  - Research Site, Vladimir
  - Research Site, Yaroslavl
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Stellenbosch
- South Korea (5):
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Jeju City
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Getafe
  - Research Site, Mérida
  - Research Site, Servilla
  - Research Site, Vigo
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Ukraine (6):
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (4):
  - Research Site, Doncaster
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Strand V, Kalunian KC, Lee KW, Seo C, Abreu G, Tummala R, Al-Mossawi H, Duncan EA, Lindholm C. Long-term effect of anifrolumab on patient-reported outcomes in systemic lupus erythematosus (TULIP-LTE): a randomised, placebo-controlled, phase 3 long-term extension trial. Lancet Rheumatol. 2025 Jul;7(7):e485-e494. doi: 10.1016/S2665-9913(25)00022-0. Epub 2025 May 2. PMID 40324450
- [Derived] Tanaka Y, Atsumi T, Okada M, Miyamura T, Ishii T, Nishiyama S, Matsumura R, Kawakami A, Hayashi N, Abreu G, Yavuz S, Lindholm C, Al-Mossawi H, Takeuchi T. The long-term safety and tolerability of anifrolumab for patients with systemic lupus erythematosus in Japan: TULIP-LTE subgroup analysis. Mod Rheumatol. 2024 Jul 6;34(4):720-731. doi: 10.1093/mr/road092. PMID 37706527
- [Derived] Kalunian KC, Furie R, Morand EF, Bruce IN, Manzi S, Tanaka Y, Winthrop K, Hupka I, Zhang LJ, Werther S, Abreu G, Hultquist M, Tummala R, Lindholm C, Al-Mossawi H. A Randomized, Placebo-Controlled Phase III Extension Trial of the Long-Term Safety and Tolerability of Anifrolumab in Active Systemic Lupus Erythematosus. Arthritis Rheumatol. 2023 Feb;75(2):253-265. doi: 10.1002/art.42392. Epub 2022 Nov 11. PMID 36369793
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00009&attachmentIdentifier=ab5090f5-1f24-42c2-b969-8f0316da65a5&fileName=D3461C00009_CSR_Synopsis_Redacted_pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This long-term extension (LTE) study was conducted at 176 study centres in 24 countries.
Pre-assignment Details: The LTE population was comprised of participants who had completed the 52-week double-blind treatment period in one of the Phase III feeder studies (D3461C00004 [NCT02446899] or D3461C00005 [NCT02446912]), met all LTE eligibility criteria, and were willing to continue into the extension study.
Groups:
- Randomised Anifrolumab 300 mg: Anifrolumab (300 mg) administered via an intravenous (IV) infusion every 4 weeks for up to 152 weeks (39 doses).
  Participants were previously administered anifrolumab (300 mg) in a feeder study.
- Placebo Feeder + Placebo LTE: Placebo administered via an IV infusion every 4 weeks for up to 152 weeks (39 doses).
  Participants were previously administered placebo in a feeder study.
- Placebo Feeder + Anifrolumab 300 mg LTE: Anifrolumab (300 mg) administered via an IV infusion every 4 weeks for up to 152 weeks (39 doses).
  Participants were previously administered placebo in a feeder study.
- Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE: Anifrolumab (300 mg) administered via an IV infusion every 4 weeks for up to 152 weeks (39 doses).
  Participants were previously administered anifrolumab (150 mg) in a feeder study.
Period: Overall Study
Arm/Group | Randomised Anifrolumab 300 mg | Placebo Feeder + Placebo LTE | Placebo Feeder + Anifrolumab 300 mg LTE | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE
Started (12 participants were enrolled but excluded due to site non-compliance or lack of source documentation.) | 257 | 112 | 111 | 67
Completed | 178 | 54 | 69 | 41
Not Completed | 79 | 58 | 42 | 26
Not completed — Adverse Event | 11 | 4 | 5 | 8
Not completed — Condition Under Investigation Improved | 1 | 0 | 0 | 0
Not completed — Condition Under Investigation Worsened | 0 | 2 | 1 | 0
Not completed — Death | 2 | 1 | 2 | 0
Not completed — Development of Study-specific Withdrawal Criteria | 1 | 0 | 0 | 1
Not completed — Failure to Meet Randomisation Criteria | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 10 | 6 | 3 | 3
Not completed — Lost to Follow-up | 5 | 6 | 3 | 1
Not completed — Severe Non-compliance to Protocol | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 38 | 29 | 20 | 12
Not completed — Missing | 1 | 0 | 0 | 0
Not completed — Due to COVID-19 Pandemic | 7 | 2 | 4 | 0
Not completed — Other - Not Due to COVID-19 Pandemic | 2 | 6 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) - LTE Study: consisted of all participants who were randomised and received at least 1 dose of investigational product in the LTE Study.
Groups:
- Randomised Anifrolumab 300 mg: Anifrolumab (300 mg) administered via an IV infusion every 4 weeks for up to 152 weeks (39 doses).
  Participants were previously administered anifrolumab (300 mg) in a feeder study.
- Total: Total of all reporting groups
Arm/Group | Randomised Anifrolumab 300 mg | Placebo Feeder + Placebo LTE | Placebo Feeder + Anifrolumab 300 mg LTE | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE | Total
Number analyzed (Participants) | 257 | 112 | 111 | 67 | 547
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 247 | 111 | 107 | 65 | 530
  >=65 years | 10 | 1 | 4 | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (11.51) | 41.4 (11.46) | 42.2 (12.24) | 42.4 (11.70) | 42.6 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 103 | 102 | 63 | 505
  Male | 20 | 9 | 9 | 4 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 173 | 77 | 70 | 45 | 365
  Black or African American | 28 | 11 | 17 | 10 | 66
  Asian | 33 | 10 | 12 | 6 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 3 | 1 | 0 | 0 | 4
  Other | 15 | 11 | 10 | 6 | 42
  Missing | 5 | 2 | 2 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 28 | 22 | 14 | 118
  Not Hispanic or Latino | 198 | 82 | 87 | 53 | 420
  Missing | 5 | 2 | 2 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Exposure-adjusted Incidence Rates (EAIRs) of Adverse Events of Special Interest (AESIs)
Description: The event rate per 100 participant years was defined as the number of participants with an event divided by the sum of exposure time during the LTE study (including follow-up) in days for all participants in the analysis set multiplied by 365.25 days/year multiplied by 100. The exposure in a time period for each participant was calculated as end of period - start of period + 1. EAIRs of AESIs are presented as event rate per 100 participant years.
  The following AESIs were pre-defined:
  * Non-opportunistic serious infections
  * Opportunistic infections
  * Anaphylaxis
  * Malignancy
  * Herpes zoster
  * Tuberculosis (TB) (including latent TB)
  * Influenza
  * Vasculitis (non-systemic lupus erythematosus [SLE])
  * Major cardiovascular events as according to the Cardiovascular Event Adjudication Committee.
Time Frame: Up to a maximum of 1114 days
Population: FAS - LTE Study: consisted of all participants who were randomised and received at least 1 dose of investigational product in the LTE Study.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Randomised Anifrolumab 300 mg | Placebo Feeder + Placebo LTE | Placebo Feeder + Anifrolumab 300 mg LTE | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE
Number analyzed (Participants) | 257 | 112 | 111 | 67
Events per 100 participant years | 11.0 | 9.6 | 12.9 | 12.5

2. Primary Outcome: EAIRs of Serious Adverse Events (SAEs)
Description: EAIRs of SAEs are presented as event rate per 100 participant years.
  An SAE was an AE occurring during any study phase that fulfils 1 or more of the following criteria:
  * Results in death
  * Is immediately life-threatening
  * Requires in-patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
  * Is a congenital abnormality or birth defect
  * Is an important medical event that may jeopardise the participant or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: Up to a maximum of 1114 days
Population: as for outcome 1
Measure: Number; unit: Events per 100 participant years
Arm/Group | Randomised Anifrolumab 300 mg | Placebo Feeder + Placebo LTE | Placebo Feeder + Anifrolumab 300 mg LTE | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE
Number analyzed (Participants) | 257 | 112 | 111 | 67
Events per 100 participant years | 8.5 | 11.2 | 10.1 | 10.7

ADVERSE EVENTS:
Time Frame: Day 1 up to until follow-up visit 2 (Week 164)
Description: FAS - LTE Study: consisted of all participants who were randomised and received at least 1 dose of investigational product in the LTE Study.
Arm/Group | Randomised Anifrolumab 300 mg | Placebo Feeder + Placebo LTE | Placebo Feeder + Anifrolumab 300 mg LTE | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE
All-Cause Mortality (participants affected / at risk) | 3/257 | 1/112 | 3/111 | 2/67
Serious Adverse Events (participants affected / at risk) | 56/257 | 27/112 | 26/111 | 14/67
Other Adverse Events (participants affected / at risk) | 195/257 | 79/112 | 81/111 | 53/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Randomised Anifrolumab 300 mg (N=257) | Placebo Feeder + Placebo LTE (N=112) | Placebo Feeder + Anifrolumab 300 mg LTE (N=111) | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE (N=67)
Herpes zoster (Infections and infestations) | 6 | 1 | 3 | 1
Pneumonia (Infections and infestations) | 6 | 2 | 3 | 3
COVID-19 (Infections and infestations) | 4/201 | 0/64 | 2/82 | 0/42 — Only participants who were ongoing in the trial at the time the COVID-19 pandemic started are included. All participants who had completed or discontinued the trial prior to the pandemic are excluded from number of participants at risk.
COVID-19 pneumonia (Infections and infestations) | 3/201 | 1/64 | 3/82 | 0/42 — Only participants who were ongoing in the trial at the time the COVID-19 pandemic started are included. All participants who had completed or discontinued the trial prior to the pandemic are excluded from number of participants at risk.
Pyelonephritis (Infections and infestations) | 3 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Ludwig angina (Infections and infestations) | 0 | 1 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 2 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Central nervous system lupus (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 6 | 6 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Incarcerated hernia (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Mucosal haemorrhage (General disorders) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomised Anifrolumab 300 mg (N=257) | Placebo Feeder + Placebo LTE (N=112) | Placebo Feeder + Anifrolumab 300 mg LTE (N=111) | Anifrolumab 150 mg Feeder + Anifrolumab 300 mg LTE (N=67)
Nasopharyngitis (Infections and infestations) | 63 | 13 | 29 | 15
Urinary tract infection (Infections and infestations) | 57 | 16 | 18 | 9
Upper respiratory tract infection (Infections and infestations) | 55 | 18 | 22 | 8
Bronchitis (Infections and infestations) | 41 | 9 | 17 | 16
Sinusitis (Infections and infestations) | 24 | 3 | 9 | 6
Pharyngitis (Infections and infestations) | 20 | 5 | 12 | 9
Oral herpes (Infections and infestations) | 19 | 6 | 6 | 0
Herpes zoster (Infections and infestations) | 16 | 6 | 12 | 10
Latent tuberculosis (Infections and infestations) | 16 | 2 | 4 | 1
Influenza (Infections and infestations) | 14 | 5 | 9 | 5
Gastroenteritis (Infections and infestations) | 7 | 7 | 13 | 3
Depression (Psychiatric disorders) | 9 | 4 | 3 | 4
Insomnia (Psychiatric disorders) | 8 | 3 | 5 | 7
Headache (Nervous system disorders) | 28 | 11 | 7 | 10
Dizziness (Nervous system disorders) | 8 | 3 | 4 | 4
Hypertension (Vascular disorders) | 13 | 4 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 4 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 18 | 6 | 8 | 5
Nausea (Gastrointestinal disorders) | 12 | 7 | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2 | 5 | 4
Constipation (Gastrointestinal disorders) | 7 | 7 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 9 | 11 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 10 | 12 | 9
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 12 | 2 | 3 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 17 | 6 | 8 | 2
Fall (Injury, poisoning and procedural complications) | 11 | 6 | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 10 | 3 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT02794285/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT02794285/SAP_001.pdf